CLINICAL TRIAL: NCT03437174
Title: Burden of Illness and Disease Associated Emergencies in Chronic Hypoparathyroidism
Brief Title: Burden of Illness in Hypoparathyroidism
Status: Completed | Type: Observational
Sponsor: University of Wuerzburg (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); University Medical Center Rostock (Other); Praxis Endokrinologie in Charlottenburg, Berlin (Unknown); Charite University, Berlin, Germany (Other); Endocrine Practice, Oldenburg, Germany (Unknown)
Responsible Party: Principal Investigator, Stefanie Hahner, Prof. Stefanie Hahner, University of Wuerzburg
Other Study IDs: BOHEME-HP
Record Dates: First submitted 2018-02-10; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Hypoparathyroidism
Keywords: Hypoparathyroidism; Parathyroid Disease; Burden of Illness; SF-36; Quality of Life
MeSH Terms: conditions — Hypoparathyroidism; Parathyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Long-term conventional treatment of chronic hypoparathyroidism does not fully restore calcium homeostasis leading to increased morbidity, emergency events and reduced subjective health status. To further investigate general morbidity, hypocalcemic events, subjective and daily life performance in patients with chronic hypoparathyroidism a disease specific questionnaire, as well as the SF-36 are handed out.

DETAILED DESCRIPTION:
Design:

In a cross-sectional trial the subjective health status and burden of illness in patients with chronic hypoparathyroidism will be evaluated by using a disease specific questionnaire as well as the SF-36.

Patients:

Patients will be recruited out of the patient population of the participating five medical centers.

Statistical Analysis:

Documentation and analysis will be performed at the Department of Medicine I, Endocrine and Diabetes Unit, University of Würzburg, Germany. Data will be documented after pseudonymisation in a data base. For further analysis data will be compared to sex- and age-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* chronic hypoparathyroidism (>12 months) under established therapy
* chronic pseudohypoparathyroidism (>12 months) under established therapy
* written informed consent

Exclusion Criteria:

* age <18 years
* no detailed documentation of hypo- or pseudohypoparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic hypo- and pseudohypoparathyroidism
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Burden of illness | 12 - 24 months
  Assessment of the burden of illness due to chronic hypoparathyroidism using a disease specific questionnaire to further investigate impairment in daily and professional life in comparison to the general German population (DEGS1, SHIP-2).

SECONDARY OUTCOMES:
Hypocalcemia | 12 - 24 months
  documentation of frequency of hypocalcemia under standard treatment
Psychological disorders | 12 - 24 months
  documentation of frequency of anxiety and depression under standard treatment
Subjective Health Status | 12-24 months
  Assessment of the subjective health status due to chronic hypoparathyroidism by Assessment of subjective health status in patients with chronic hypoparathyroidism

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Hahner, MD, Principal Investigator — University Hospital Wuerzburg
Locations (5):
- Germany (5):
  - Endokrinologie in Charlottenburg, Berlin
  - Charite Berlin, Berlin
  - Ludwig-Maximilians-Universität, Munich
  - University Hospital Rostock, Rostock
  - Dept. of Endocrinology and Diabetology, Dept. of Medicine I, University Hospital Wuerzburg, Würzburg

REFERENCES:
- [Background] Arlt W, Fremerey C, Callies F, Reincke M, Schneider P, Timmermann W, Allolio B. Well-being, mood and calcium homeostasis in patients with hypoparathyroidism receiving standard treatment with calcium and vitamin D. Eur J Endocrinol. 2002 Feb;146(2):215-22. doi: 10.1530/eje.0.1460215. PMID 11834431
- [Background] Hadker N, Egan J, Sanders J, Lagast H, Clarke BL. Understanding the burden of illness associated with hypoparathyroidism reported among patients in the PARADOX study. Endocr Pract. 2014 Jul;20(7):671-9. doi: 10.4158/EP13328.OR. PMID 24449664